CLINICAL TRIAL: NCT05685862
Title: Laser Speckle Contrast Imaging, Surgical Eye and Indocyanine Green Fluorescence Imaging for Perfusion Assessment of the Gastric Conduit
Brief Title: Laser Speckle Contrast Imaging, Surgical Eye & ICG Fluorescence Imaging for Perfusion Assessment of the Gastric Conduit
Acronym: CONDOR-I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Frisius Medisch Centrum (Other)
Collaborators: University of Groningen (Other); LIMIS Development (Unknown)
Responsible Party: Principal Investigator, E.C. Boerma, Dr., Frisius Medisch Centrum
Other Study IDs: NL81217.099.22
Record Dates: First submitted 2022-09-13; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Oesophageal Cancer
Keywords: Laser Speckle Contrast Imaging; LSCI; gastric conduit; oesophageal cancer; ICG; fluorescence
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: All patients eligible to participate in this study.
  Interventions: Device: Laser Speckle Contrast Imaging using the PerfusiX-Imaging device

INTERVENTIONS:
Device: Laser Speckle Contrast Imaging using the PerfusiX-Imaging device — Patient will undergo the standard-of-care gastric conduit procedure and in addition, peroperative Laser Speckle Contrast Imaging of the gastric conduit and eosophagus will be performed.

SUMMARY:
Rationale Globally, esophageal cancer is the seventh most common cancer type, with over half a million cases reported in 2020. The survival of gastroesophageal cancer is poor and the prognosis is primarily determined by the possibilities for curative treatment. After resection of part of the esophagus and cardia, the reconstruction of the esophagus is performed with a gastric conduit where an anastomosis is made with the proximal esophageal stump. Globally, a Minimally invasive Esophagectomy (MIE) has a high morbidity rate and a mortality rate ranging up to 5% as a result of the procedure. One of the most feared complications is an anastomotic leakage (AL) with a rate of around 12.5% and a mortality rate of around 15%. AL is associated with prolonged hospital stay and increased re-operation rates. It is generally accepted that impaired blood flow of the gastric conduit is the most important cause of AL. The surgical procedure of an esophagectomy and reconstruction inherently compromises the blood supply of the gastric conduit. However other than the surgical eye, there is no gold standard in assessing this. Surgeons generally look for traditional indicators of tissue viability such as pulsating vessels, bleeding of the resected edges, tissue color and intestinal motility. However, an objective indication of the tissue perfusion is still lacking, implying the clinical need for one.

Objectives In this trial the investigators will study the utility of PerfusiX-Imaging for perfusion assessment of the gastric conduit in comparison with the standard of care.

Study design The current study is a prospective, observational single-center study in the Medical Center Leeuwarden.

Study population A total of 30 patients undergoing an esophageal resection will be included. Patient related study procedures All patients will undergo the standard-of-care program which includes perfusion assessment by the surgical eye and ICG-fluorescence imaging. In addition to this standard-of-care, 2D-perfusion maps will be generated from images taken with PerfusiX-Imaging (LIMIS Development BV, Leeuwarden, The Netherlands) in combination with a standard surgical laparoscope. Not related to the patient, the PerfusiX-Imaging images will be shown to the surgeon postoperatively and peroperative questionnaires will be filled regarding the standard-of-care perfusion assessment.

Study parameters/endpoints Due to the explorative character of this study, there is no formal hierarchy in the respective endpoints of this study. In this, all endpoints will add to the overall assessment of the feasibility of the PerfusiX-imaging derived visual feedback. The investigators will look at the percentage of operating surgeons that indicated no change in location of the anastomosis or operating plan based on the additional PerfusiX-Imaging. The percentage of the non-involved surgeons that indicated no change in location of the anastomosis or operating plan based on the additional PerfusiX-Imaging. And the homogeneity of the change in location between non-involved surgeons for individual patients will be analyzed in order to get a sense for the subjectivity of the interpretation of the images.

The investigators will also compare the additional PerfusiX-Imaging derived visual feedback to the standard of care by looking at the homogeneity in location of the watershed area between PerfusiX-Imaging, ICG-fluorescence and based on visual assessment by the surgical eye. The difference in the location of watershed area between PerfusiX-Imaging and ICG-fluorescence or based on visual assessment.

In order to get a sense of the scale of the indicated change in location of the anastomosis the investigators will look at the estimated change in location of the anastomosis of the gastric conduit/ the esophageal stump in centimeters by the operating surgeon. The estimated change in location of the anastomosis of the gastric conduit/ the esophageal stump in centimeters by non-involved surgeons. Lastly, the investigators will compare the change in the location of the anastomosis by non-involved surgeons in comparison to the operating surgeon; Burden, risk and benefit to participation Burden Not applicable. Risks Not applicable. Benefit Not applicable.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE 1.2 Perfusion defects associated with anastomotic leakage It is generally accepted that impaired blood flow of the gastric conduit is the most important cause of AL. The surgical procedure of an esophagectomy and reconstruction inherently compromises the blood supply of the gastric conduit. This is mainly due to the fact that the blood supply of the gastric conduit is solely dependent on the right gastroepiploic artery. Good condition and length of this artery and the microvasculature of the gastric wall is thus of utmost importance. Unfortunately, the cardiovascular condition of the patient is affected by many uncontrollable risk factors such as diabetes, smoking, hypertension but also neo-adjuvant chemoradiotherapy. Surgeons are well aware of the risks of poor perfusion of the gastric conduit, and the subsequent AL. However other than the clinical experience / surgical eye, there is no validated method for assessing this. Surgeons generally look for traditional indicators of tissue viability such as pulsating vessels, bleeding of the resected edges, tissue color and intestinal motility. However, an objective estimation of the tissue perfusion is still lacking, implying the clinical need for one. In this study the investigators will study the utility of laser speckle contrast imaging (LSCI) for this purpose. The results will be compared to the current standard-of-care; indocyanine green (ICG) imaging and the surgical eye.

   1.3 Laser speckle contrast imaging About the perfusion imaging technique; LSCI. The first biomedical application of LSCI was reported in the 1981 by Fercher and Biers. The proposed technique from Fercher and Briers was non-real-time and had its practical limitations due to the use of non-digital systems which impeded the clinical use. The first real speed increase to quasi real-time image acquisition and processing happened in the nineties with the introduction of digital photography. Generally, the components required are a low-powered laser diode, a diffuser, a digital camera and processing software (Figure 1). Other names for the same principle as LSCI are laser speckle imaging (LSI), laser speckle perfusion imaging (LSPI) and laser speckle contrast analysis (LASCA) as it was named by the first users.

   1.4 The basic principle of laser speckle contrast imaging Speckle patterns are the random interference patterns that arise when coherent light is backscattered by a scattering medium such as biological tissue. The slightly different optical pathlengths cause the waves to reach the observer at random mutual phases, resulting in bright and dark spots respectively9. The speckle image is built up of static and dynamic speckles. Static speckles are speckles that do not change over time whereas dynamic speckles do change over time due to the optical Doppler effect. The dynamic speckles contain information about movement of the object, or motion of particles within the object.

   In order to be able to detect a change in the speckle pattern, the exposure time of the camera must be of the order of the speckle decorrelation time, causing a blurring of the recorded speckle pattern. It is this blurring that is used to calculate the speckle contrast K using the following formula 1.

   K=σ/(<I>) (1) Where σ is the standard deviation of the intensity I over the mean intensity <I> calculated over a window in space or time. Spatial contrast uses an area of multiple pixels in one frame as can be seen in the bottom left corner of Figure 2. A window size of 5 x 5 or 7 x 7 pixels has been suggested for optimal results. As spatial contrast decreases the spatial resolution, however, this method does have a high temporal resolution. Temporal LSCI uses the same pixel in multiple frames to calculate the contrast in a time window as can be seen in the top right corner of Figure 2. Temporal contrast has a high spatial resolution and low temporal resolution. For spatial contrast this is vice versa and hence, it can be beneficial if combined into a so-called spatio-temporal contrast. The choice of resolution should be based on the need for a high temporal or spatial resolution.

   If the exposure time of the detector is shorter than the intensity fluctuation time of the speckles, the standard deviation σ is equal to the mean intensity <I> which theoretically results in a contrast value of K=1. If there is movement present and the exposure time of the detector is of the order of, or longer than the fluctuation time, the picture will be blurred meaning that the standard deviation σ will be small compared to the mean intensity <I> which results in a loss of contrast, hence 0≥K<1.

   1.5 Standard-of-care: Indocyanine green fluorescence imaging The use of ICG is standard-of-care in the MCL and ICG and its application for perfusion assessment are CE-certified and will be used as approved. The ICG procedure described in this protocol is according to the standard MCL ICG protocol (See addendum K6.16). Indocyanine green is a water-soluble anionic amphiphilic tricarbocyanine dye with a molecular weight of 774.96 Da. It becomes completely and permanently fixed to plasma proteins once in the bloodstream, and circulates in the intravascular compartment only. This may allow for the blood flow of the gastric conduit to be visualized. This dye can be injected into the human bloodstream with practically no adverse effects. It becomes fluorescent upon excitation by a laser beam or by light with a wavelength in the near infra-red (NIR) spectrum (approximately 820 nm). This dye was first approved for clinical use in 1956 and is now, next to methylene blue the only clinically food and drug administration (FDA) and European Medicines Agency (EMA) approved fluorescent dye. Twenty-five mg of ICG will be dissolved in 10mL sterile water (2.5mg/mL). The ICG fluorescence will be imaged using the Olympus Viscera ELITE II infrared imaging system.

   1.6 Rationale for the CONDOR-I study The current intraoperative assessment of perfusion around the site for the anastomosis is based on subjective clinical indicators of intestinal viability, i.e. the surgeon's eye and ICG-fluorescence imaging. As indicated by others12 there is a need for a gold standard in determining the state of microcirculation. This method should be suitable for laparoscopic use, robust and preferably non-invasive. Our hypothesis is that PerfusiX-Imaging could be this method. By comparing PerfusiX-Imaging to the current standard-of-care perfusion assessment (i.e., ICG-fluorescence and the surgical eye), the most optimal method for real-time feedback can be obtained and used for clinical decision-making during surgery, which might be beneficial to the patient. This benefit can be the result of two actions; (1) repositioning of the location of the anastomosis or (2) a change in operating plan. Repositioning the location of the anastomosis is helpful when this is repositioned in a better perfused area. A change in operating plan could be a Roux-y reconstruction or a colon interponate instead of a gastric tube reconstruction. In this prospective observational feasibility study, the investigators aim to determine whether the added clinical value and whether the operating plan would have changed, based on additional PerfusiX-imaging derived visual feedback.
2. OBJECTIVES 2.1 Primary objectives Due to the explorative character of this study, there is no formal hierarchy in the respective objectives of this study. In this, all objectives will add to the overall assessment of the feasibility of the PerfusiX-imaging derived visual feedback.

   * To determine whether operating surgeons, based on additional PerfusiX-imaging derived visual feedback, in hindsight would have changed the location of the anastomosis or operating plan.
   * To determine whether non-involved surgeons, based on additional PerfusiX-imaging derived visual feedback, in hindsight would have changed the location of the anastomosis or operating plan.
   * To determine the change in location of the anastomosis (if indicated that the anastomosis would be relocated) by the operating surgeon (in centimeters).
   * To determine the change in location of the anastomosis (if indicated that the anastomosis would be relocated) by non-involved surgeons (in centimeters).
   * To determine the homogeneity of the decision to change the location between the non-operating surgeons for individual patients.
   * To determine if there is overlap between the location of the watershed area as indicated by PerfusiX-Imaging, the ICG-fluorescence, and the surgical eye.

2.2 Secondary objectives Not applicable. 3. STUDY DESIGN The current study is a prospective, observational single-center study in the Medical Center Leeuwarden. A total of 30 patients undergoing an esophageal resection will be included (see section 4 'Study population'). Patients will - after written informed consent - undergo the regular standard-of-care program (i.e. perfusion assessment by means of the surgical eye and ICG-fluorescence imaging). In addition to this standard-of-care, 2D-perfusion maps will be generated from images taken with PerfusiX-Imaging (LIMIS Development BV, Leeuwarden, The Netherlands) in combination with a standard, unmodified surgical laparoscope and video system (EndoEye, Olympus Medical, Hamburg, Germany). The images will be shown to the surgeon postoperatively and per operative questionnaires will be filled by the surgeon. A detailed description of the safety aspects, application and specification of these devices can be found in section 6 and 7. A detailed description of the imaging protocol can be found in section 8.

4 STUDY POPULATION 4.1 Population All included patients meeting the eligibility criteria and scheduled to undergo esophageal resection.

4.2 Inclusion criteria

In order to be eligible to participate in this study, the subject must meet all following criteria:

* Scheduled to undergo esophageal resection;
* Age 18 years or older;
* Written informed consent; 4.3 Exclusion criteria
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent; 4.4 Sample size calculation For this explorative study, no formal sample size calculation was performed. A total of 30 patients total is deemed sufficient by experts to determine the effect of PerfusiX-Imaging on the surgeon's clinical decision making. With this number of patients, it is likely for some patients to develop anastomotic leakage. There is no consensus in the literature regarding the incidence of AL in esophageal surgery. Numbers range between 8.5% and 24.5%.13-17 Assuming a 12.5% chance of anastomotic leakage, a total of 4 patients out of 30 patients will develop anastomotic leakage. Data on patients developing AL could be useful for future studies. For the assessments by the non-operating surgeons, at least 5 non-involved surgeons will assess each patient case. Results of this study will be used for a power size calculation for a possible subsequent intervention study in order to determine the effectiveness of PerfusiX-Imaging as a tool to prevent AL.

  5 TREATMENT OF SUBJECTS 5.1 Investigational product/treatment The investigational medical device is a medical imaging device that uses LSCI as a technology to image perfusion of the gastric conduit. This technology is referred to in literature as laser speckle contrast imaging, laser speckle contrast analyses or laser speckle perfusion imaging. There is no change in treatment for the patients included in this study. As ICG-fluorescence imaging and the surgical eye are used for the assessment of the gastric conduit perfusion. The ICG-fluorescence device (Olympus, Hamburg, Germany) is a CE-certified device that is used on label.

5.2 Use over co-intervention (if applicable) Not applicable. 5.3 Escape medication (if applicable) Not applicable.

6 INVESTIGATIONAL DEVICE 6.1.2 Positioning in the operating room Positioning of the research set-up is outside the sterile zone of the operating room (OR). The fiber optic cable between the white light source and the laparoscope will be replaced by a connection between the white light source and the investigational medical device.

6.2 Summary of findings from non-clinical studies Not applicable. 6.3 Summary of findings from clinical studies A feasibility study has been published recently in the international scientific journal "Biomedical Optics Express" which used a similar setup as the current investigational device. In the first work, the feasibility of LSCI as a tool for imaging perfusion is studied21. This work is proof that the investigational medical device is capable of measuring perfusion. An experimental setup was developed using a green 532nm and red 680nm laser and commercially available laparoscopic video systems. Vascular occlusion tests (VOT) performed on the large intestines and the nail fold were analyzed using custom software and were compared with published data. Ten (n=10) subjects undergoing colonic resections were included in a two-center study and of ten (n=10) healthy volunteers participated in the VOT nail fold experiment. The 532nm laser showed significant differences of 90.46 ± 3.78% (p<0.0001) and 81.08 ± 4.22% (p<0.0001) during occlusion, 107.51 ± 5.56% (p=0.005) and 108.53 ± 8.51% (p=0.148) during reperfusion compared to the baseline for the intestines and nail fold respectively. Also, the post-occlusion plateau differed significantly from baseline, 99.64 ± 6.11% (p=0.86), on the nail fold. The 680nm laser showed a significant decrease, 81.08 ± 4.22% (p<0.0001), during occlusion of the nail fold and did not show significant differences during the other phases. This two-center study with ten (n=10) subjects undergoing a colonic resection illustrates that laser speckle contrast imaging is capable of identifying ischemic areas on the large intestine in a standard laparoscopic setup with a measured flow decrease of up to 10% compared to baseline level. Other clinical applications of LSCI can be found in this review 22.

Additionally, Milstein et al. have performed LSCI measurements one the gastric conduit following esophagectomy with positive results. A notable difference between this study and the study by Milstein et al. is that the investigators will use a laparoscopic LSCI device as to compared to an open surgical device23.

6.4 Summary of know and potential risks and benefits See IMDD (Version 1.1, November 2020, section 5) for a summary of known and potential risks and benefits of laparoscopic LSCI.

7 NON-INVESTIGATIONAL PRODUCT 7.1 Name and description of non-investigation product(s) 7.1.1 Olympus surgical OTV-S300 video processor The OTV-S300 is an all-in-one 2D/3D processor and light source for laparoscopic surgeries. It is capable of both 2D and 3D observation packed in a compact system for a simplified workflow. It has an LCD touch panel that allows for presets for easy preparation and maintenance. It has an LED light source which produces good natural color reproduction with the combination of enhanced imaging processes. It has spectral light observation with narrowband imaging and two modes of IR-observation.

8 METHODS 8.1 Study parameters/endpoints 8.1.1 Study parameter/endpoint Due to the explorative character of this study, there is no formal hierarchy in the respective endpoints of this study. In this, all endpoints will add to the overall assessment of the feasibility of the PerfusiX-imaging derived visual feedback.

The investigators will look at the percentage of operating surgeons that indicated no change in location of the anastomosis or operating plan based on the additional PerfusiX-Imaging. The percentage of the non-involved surgeons that indicated no change in location of the anastomosis or operating plan based on the additional PerfusiX-Imaging. And the homogeneity of the change in location between non-involved surgeons for individual patients will be analyzed in order to get a sense for the subjectivity of the interpretation of the images.

The investigators will also compare the additional PerfusiX-Imaging derived visual feedback to the standard of care by looking at the homogeneity in location of the watershed area between PerfusiX-Imaging, ICG-fluorescence and based on visual assessment by the surgical eye. The difference in the location of watershed area between PerfusiX-Imaging and ICG-fluorescence or based on visual assessment.

In order to get a sense of the scale of the indicated change in location of the anastomosis the investigators will look at the estimated change in location of the anastomosis of the gastric conduit/ the esophageal stump in centimeters by the operating surgeon. The estimated change in location of the anastomosis of the gastric conduit/ the esophageal stump in centimeters by non-involved surgeons. Lastly, the investigators will compare the change in the location of the anastomosis by non-involved surgeons in comparison to the operating surgeon;

The overlap in location of the watershed area between the modalities (LSCI, ICG-fluorescence and the surgical eye) will be determined to assess clinical applicability of LSCI in esophagus-surgery.

8.1.2 Other study parameters/endpoints (if applicable)

- Not applicable 8.2 Randomization, blinding and treatment allocation The current study is a non-randomized, non-blinded, prospective, single-center in which all patients are scheduled to undergo a surgical procedure according to standard care. There is no difference in therapeutic procedure among included patients.

8.3 Study procedures 8.3.1 Inclusion procedure Potential eligible patients are identified by their treating physician (in Dutch: hoofdbehandelaar). The treating physician will assess eligibility by checking in- and exclusion criteria based on the available data (according to paragraph 4.2 and 4.3). If a patient is found to be eligible to participate in the study, he or she will receive oral information about the study during a standard clinic visit, several weeks prior to surgical procedure. In addition, he or she will receive written study information (together with the standard information) and is asked to consider participation. The patients will be informed about the aim of the study, the procedures and associated risks before enrolment into the study. Also, patients will be informed as to the strict confidentiality of their data.

Two weeks after receiving the information about the study, patients can inform their treating physician or the secretary staff of the Chirurgie MCL in person, by phone, mail or e-mail to confirm that they are willing to participate in this study. When patients agree to participate, signed written informed consent is obtained. For more specified information about informed consent, see chapter 11.2.

8.3.2 Image acquisition protocol The patient will be treated according to treatment plan as was established by the treating physician. The surgical procedure is executed as is deemed appropriate by the surgeon. The image acquisition protocol is executed in both the thoracic and the abdominal phase of the surgery. There will be three imaging moments where the investigators will image using PerfusiX-Imaging. Additionally, the standard-of-care ICG-imaging and visual assessment will be noted based on the surgeons' judgement. The three imaging moments are (1) baseline during the abdominal phase (2) After making the gastric conduit and (3) imaging of the tip of the gastric conduit and esophageal stump before making the anastomosis in the thoracic phase. This is represented in the table below.

The LSCI images will NOT be shown during surgery to any surgeon. 8.3.3 Perioperative visual assessment (operating surgeon) During the three measuring moments the on-site investigator will ask the surgeon to fill out the short peroperative questionnaire based on the visual inspection and ICG-fluorescence imaging of the state of perfusion of the tissue.

8.3.4 Postoperative indication of change in clinical decision making (operating surgeon) The investigators will show the images to the operating surgeon directly after surgery and ask him/her whether he/she would change the location of the anastomosis or operating plan based on the additional PerfusiX-Imaging derived visual feedback.

8.3.5 Postoperative change in clinical decision making (non-involved surgeon) After all inclusions the investigator will ask other, non-involved surgeons to determine the endpoints of this study concerning clinical decision making. The investigators will show the images to the non-involved surgeons and ask them whether they would change the location of the anastomosis based on the additional PerfusiX-Imaging derived visual feedback. In this, each assessor (at least) 5 surgeons will first make his/her own decision. Thereafter, consensus can be reached for inconclusive cases.

8.3.6 Anastomotic leakage check Minimally 30 days after the imaging procedure, the investigators will examine the patients electronic patient file to check if the patient was diagnosed by the treating surgeon with anastomotic leakage.

8.4 Withdrawal of individual subjects Subjects can leave the study at any time prior to surgery for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons.

8.4.1 Specific criteria for withdrawal (if applicable) Subjects will be withdrawn from the study when no surgery will be performed. 8.5 Replacement of individual subjects after withdrawal Patient who are withdrawn will be replaced in this study. 8.6 Follow-up of subjects withdrawn from treatment Not applicable. 8.7 Premature termination of the study 8.7.1 Termination based on safety aspects Not applicable 8.7.2 Termination based on other aspects The study will be suspended based on urgent medical or ethical considerations as decided by the principal investigators. In case of termination of the study, the institution, regulatory authorities, CCMO and the METC of the study center will be informed.

9 SAFETY MONITORING 9.1 Temporary halt for reasons of subject safety In accordance to section 10, subsection 4 of the WMO, the sponsor will suspend the study if there is sufficient ground that continuation of the study will jeopardize subject health or safety. The sponsor will notify the accredited METC without undue delay of a temporary halt including the reason for such an action. The study will be suspended pending a further positive decision by the accredited METC. The investigator will take care that all subjects are kept informed.

9.2 AEs, SAEs 9.2.1 Adverse events (AEs) Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the investigational product. All adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded.

9.2.2 Serious adverse events (SAEs) A serious adverse event is any untoward medical occurrence or effect that

* results in death;
* is life threatening (at the time of the event);
* requires hospitalization or prolongation of existing inpatients' hospitalization;
* results in persistent or significant disability or incapacity;
* is a congenital anomaly or birth defect; or
* any other important medical event that did not result in any of the outcomes listed above due to medical or surgical intervention but could have been based upon appropriate judgement by the investigator.

An elective hospital admission will not be considered as a serious adverse event.

The sponsor will report the SAEs through the web portal ToetsingOnline to the accredited METC that approved the protocol, within seven days of first knowledge for SAEs that result in death or are life threatening followed by a period of maximum of eight days to complete the initial preliminary report. All other SAEs will be reported within a period of maximum 15 days after the sponsor has first knowledge of the serious adverse events.

9.2.3 Suspected unexpected serious adverse reactions (SUSARs) Not applicable. 9.3 Annual safety report Not applicable. 9.4 Follow-up of adverse events All AEs that are related to the investigational medical product will be followed until they have abated, or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated, and/or referral to the general physician or a medical specialist. SAEs need to be reported till end of study within the Netherlands, as defined in the protocol.

9.5 Data Safety Monitoring Board (DSMB) An independent external Data Safety Monitoring Board of experts will not be instituted.

10 STATISTICAL ANALYSIS The overall aim of this study is to see if the use of additional PerfusiX-Imaging derived visual feedback alters the determination the optimal location of the anastomosis compared to the standard of care. For this the investigators determine the percentage of surgeons that indicate no change in surgical plan based on the additional PerfusiX-Imaging derived visual feedback. Descriptive statistics will include measurements of distribution: (geometric) means with standard deviation; medians with range; frequencies with 95% confidence interval.

11 ETHICAL CONSIDERATIONS 11.1 Regulation statement The study will be conducted according to the principles of the Declaration of Helsinki (Fortaleza, Brazil, 2013 amendment) and in accordance with the Medical Research Involving Human Subjects Act (WMO) and other guidelines, regulations and Acts. The protocol has been written and the study will be conducted according to the ICH Harmonized Tripartite Guideline for Good Clinical Practice. The protocol will be approved by the Local, Regional or National Ethics Committees.

11.2 Recruitment and consent Recruitment is done by the operating surgeon of the patient. All subjects are informed and asked for their consent. The minimal time between first appointment with doctor and surgery is 2 weeks, what results in a minimal time of 2 weeks for consideration.

Written informed consent must be obtained for all patients included in the study before they are registered in the study. Patients must be given adequate opportunity to read the information and enquire about details of the study before consent is given. This implies that the written informed consent form will be signed and personally dated by the patient. The informed consent statement will be signed and dated by the investigator afterwards and the patient will receive a copy. The general physician of each patient will be informed about the enrollment of the patient to the study.

11.3 Objection by minors or incapacitated subjects (if applicable) Not applicable. 11.4 Benefits and risk assessment, group relatedness All patients included in the study will be treated comparable with patients not included in the study. The difference between non-included and included patients is prolonged operating time. Prolonged operating time can increase the risk for patients, (e.g. infection (although this is rather minimal for laparoscopic surgery) and prolonged narcosis. The results do not immediately benefit the patients included in this study, but could help future patients to improve patient outcome.

11.5 Compensation for injury

The sponsor/investigator has a liability insurance which is in accordance with article 7 of the WMO. The sponsor (also) has insurance which is in accordance with the legal requirements in the Netherlands (Article 7 WMO). This insurance provides cover for damage to research subjects through injury or death caused by the study. The total amounts of insurance are as follows:

1. A maximum of €650.000 (i.e. six hundred and fifty thousand euros) for death or injury for each subject who participates in this current research;
2. A maximum of €5.000.000 (i.e. five million five hundred thousand euros) for death or injury for all subjects who participate in this current research;
3. A maximum of €7.500.000 (i.e. seven million five hundred thousand euros) for the total damage that becomes apparent at the study participant in research which was conducted by the Medical Center Leeuwarden. Act in each year of insurance coverage.

The insurance applies to the damage that becomes apparent during the study or within 4 years after the end of the study.

11.6 Incentives (if applicable) Not applicable.

12 ADMINISTRATIVE ASPECTS, MONITORING AND PUBLICATION 12.1 Handling and storage of data and documents Data of patients will be handled confidentially and a coded identification number (study protocol number 'CONDOR' followed by number of inclusion (for example CONDOR01) will be used to link the data to the specific patient. Data that can be linked to a specific patient will be stored separately. The principal investigator safeguards the key to the code. The handling of the personal data complies with the EU General Data Protection Regulation and the Dutch Act on Implementation of the General Data Protection Regulation (in Dutch: Uitvoeringswet AVG, UAVG)). These data will be stored at the specific site for at least fifteen years.

For software adjustments a software engineer from ZiuZ Research BV can have access to only the images. All images are coded with the patient number, location of image, type of image, with/without surgical clip and only accessible by a password. For example:

"60-D-LSCI-SCY" This describes an image of patient 60, distal end, LSCI image, surgical clip is placed.

12.3 Amendments

Amendments are changes made to the research after a favorable opinion by the accredited METC has been given. All amendments will be notified to the METC that gave a favorable opinion. A 'substantial amendment' is defined as an amendment to the terms of the METC application, or to the protocol or any other supporting documentation, that is likely to affect to a significant degree:

* the safety or physical or mental integrity of the subjects of the trial;
* the scientific value of the trial;
* the conduct or management of the trial; or
* the quality or safety of any intervention used in the trial. All substantial amendments will be notified to the METC and to the competent authority. Non-substantial amendments will not be notified to the accredited METC and the competent authority, but will be recorded and filed by the sponsor.

12.4 Annual progress report The sponsor/investigator will submit a summary of the progress of the trial to the accredited METC once a year. Information will be provided on the date of inclusion of the first subject, numbers of subjects included and numbers of subjects that have completed the trial, serious adverse events/ serious adverse reactions, other problems, and amendments.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo esophageal resection;
* Age 18 years or older;
* Written informed consent;

Exclusion Criteria:

- Medical or psychiatric conditions that compromise the patient's ability to give informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting the eligibility criteria and scheduled to undergo esophageal resection in the Medical Center Leeuwarden.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Indication of change in location or operating plan of anastomosis by operating surgeon based on PerfusiX-Imaging in comparison to standard-of-care | 1 day
  - Number of operating surgeons to indicate a change in location of anastomosis (Yes/no, %, with 95% confidence interval)
Indication of change in location or operating plan of anastomosis non-involved surgeon based on PerfusiX-Imaging in comparison to standard-of-care | 1 day
  - Number of non-involved surgeons to indicate a change in location of anastomosis (Yes/no, %, with 95% confidence interval)
Difference in location of watershed area | 1 day
  - Difference in location of watershed area in centimeters between PerfusiX, ICG-fluorescence and surgical eye (Means with standard deviation, median with range)
Estimated direction of change in location by operating surgeon in comparison to standard-of-care | 1 day
  - Proximal or medial direction of change (Yes/no, %, with 95% confidence interval)
Estimated distance of change in location by operating surgeon in comparison to standard-of-care | 1 day
  - Change in location of anastomosis in centimeters (Means with standard deviation, median with range)
Estimated direction of change in location by non-involved surgeon in comparison to standard-of-care | 1 week
  - Proximal or medial direction of change (Yes/no, %)
Estimated distance of change in location by non-involved surgeon in comparison to standard-of-care | 1 week
  - Change in location of anastomosis in centimeters (Means with standard deviation, median with range)
Indication of change in direction of anastomosis non-involved surgeon based on PerfusiX-Imaging in comparison to standard-of-care | 1 week
  - Proximal or medial direction of change (Yes/no, %, with 95% confidence interval)
Indication of change in centimeters of anastomosis non-involved surgeon based on PerfusiX-Imaging in comparison to standard-of-care | 1 week
  - Change in location of anastomosis in centimeters (Means with standard deviation, median with range)
Development of anastomotic leakage | 3 months from the moment of surgery
  - Number of patients developing AL (Percentage, %, with 95% confidence interval)
Characteristics of anastomotic leakage if present | 3 months from the moment of surgery
  - AL characteristics (localization, tumor type, type of hemicolectomy, diagnosed with, treatment)
Extra time taken for imaging | 1 day, during surgery.
  - Extra time taken for imaging protocol in seconds (Means with standard deviation, median with range)

CONTACTS AND LOCATIONS:
Overall Officials: E.C. Boerma, MD/PhD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Center Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luketich JD, Pennathur A, Awais O, Levy RM, Keeley S, Shende M, Christie NA, Weksler B, Landreneau RJ, Abbas G, Schuchert MJ, Nason KS. Outcomes after minimally invasive esophagectomy: review of over 1000 patients. Ann Surg. 2012 Jul;256(1):95-103. doi: 10.1097/SLA.0b013e3182590603. PMID 22668811
- [Background] Biere SS, van Berge Henegouwen MI, Maas KW, Bonavina L, Rosman C, Garcia JR, Gisbertz SS, Klinkenbijl JH, Hollmann MW, de Lange ES, Bonjer HJ, van der Peet DL, Cuesta MA. Minimally invasive versus open oesophagectomy for patients with oesophageal cancer: a multicentre, open-label, randomised controlled trial. Lancet. 2012 May 19;379(9829):1887-92. doi: 10.1016/S0140-6736(12)60516-9. Epub 2012 May 1. PMID 22552194
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Kassis ES, Kosinski AS, Ross P Jr, Koppes KE, Donahue JM, Daniel VC. Predictors of anastomotic leak after esophagectomy: an analysis of the society of thoracic surgeons general thoracic database. Ann Thorac Surg. 2013 Dec;96(6):1919-26. doi: 10.1016/j.athoracsur.2013.07.119. Epub 2013 Sep 24. PMID 24075499
- [Background] van Heijl M, Omloo JM, van Berge Henegouwen MI, Hoekstra OS, Boellaard R, Bossuyt PM, Busch OR, Tilanus HW, Hulshof MC, van der Gaast A, Nieuwenhuijzen GA, Bonenkamp HJ, Plukker JT, Cuesta MA, Ten Kate FJ, Pruim J, van Dekken H, Bergman JJ, Sloof GW, van Lanschot JJ. Fluorodeoxyglucose positron emission tomography for evaluating early response during neoadjuvant chemoradiotherapy in patients with potentially curable esophageal cancer. Ann Surg. 2011 Jan;253(1):56-63. doi: 10.1097/SLA.0b013e3181f66596. PMID 21233607
- [Background] Pham TH, Perry KA, Enestvedt CK, Gareau D, Dolan JP, Sheppard BC, Jacques SL, Hunter JG. Decreased conduit perfusion measured by spectroscopy is associated with anastomotic complications. Ann Thorac Surg. 2011 Feb;91(2):380-5. doi: 10.1016/j.athoracsur.2010.10.006. PMID 21256274
- [Background] Briers JD, Fercher AF. Retinal blood-flow visualization by means of laser speckle photography. Invest Ophthalmol Vis Sci. 1982 Feb;22(2):255-9. PMID 7056639
- [Background] Draijer M, Hondebrink E, van Leeuwen T, Steenbergen W. Review of laser speckle contrast techniques for visualizing tissue perfusion. Lasers Med Sci. 2009 Jul;24(4):639-51. doi: 10.1007/s10103-008-0626-3. Epub 2008 Dec 3. PMID 19050826
- [Background] Boas DA, Dunn AK. Laser speckle contrast imaging in biomedical optics. J Biomed Opt. 2010 Jan-Feb;15(1):011109. doi: 10.1117/1.3285504. PMID 20210435
- [Background] Karliczek A, Harlaar NJ, Zeebregts CJ, Wiggers T, Baas PC, van Dam GM. Surgeons lack predictive accuracy for anastomotic leakage in gastrointestinal surgery. Int J Colorectal Dis. 2009 May;24(5):569-76. doi: 10.1007/s00384-009-0658-6. Epub 2009 Feb 17. PMID 19221768
- [Background] Wei HJ, Xing D, Lu JJ, Gu HM, Wu GY, Jin Y. Determination of optical properties of normal and adenomatous human colon tissues in vitro using integrating sphere techniques. World J Gastroenterol. 2005 Apr 28;11(16):2413-9. doi: 10.3748/wjg.v11.i16.2413. PMID 15832410
- [Background] Chu M, Vishwanath K, Klose AD, Dehghani H. Light transport in biological tissue using three-dimensional frequency-domain simplified spherical harmonics equations. Phys Med Biol. 2009 Apr 21;54(8):2493-509. doi: 10.1088/0031-9155/54/8/016. Epub 2009 Apr 1. PMID 19336841
- [Background] Wei HJ, Xing D, Wu GY, Gu HM, Lu JJ, Jin Y, Li XY. Differences in optical properties between healthy and pathological human colon tissues using a Ti:sapphire laser: an in vitro study using the Monte Carlo inversion technique. J Biomed Opt. 2005 Jul-Aug;10(4):44022. doi: 10.1117/1.1990125. PMID 16178655
- [Background] Hidovic-Rowe D, Claridge E. Modelling and validation of spectral reflectance for the colon. Phys Med Biol. 2005 Mar 21;50(6):1071-93. doi: 10.1088/0031-9155/50/6/003. Epub 2005 Feb 23. PMID 15798309
- [Background] Heeman W, Dijkstra K, Hoff C, Koopal S, Pierie JP, Bouma H, Boerma EC. Application of laser speckle contrast imaging in laparoscopic surgery. Biomed Opt Express. 2019 Mar 25;10(4):2010-2019. doi: 10.1364/BOE.10.002010. eCollection 2019 Apr 1. PMID 31086715
- [Background] Heeman W, Steenbergen W, van Dam G, Boerma EC. Clinical applications of laser speckle contrast imaging: a review. J Biomed Opt. 2019 Aug;24(8):1-11. doi: 10.1117/1.JBO.24.8.080901. PMID 31385481
- [Background] Milstein DMJ, Ince C, Gisbertz SS, Boateng KB, Geerts BF, Hollmann MW, van Berge Henegouwen MI, Veelo DP. Laser speckle contrast imaging identifies ischemic areas on gastric tube reconstructions following esophagectomy. Medicine (Baltimore). 2016 Jun;95(25):e3875. doi: 10.1097/MD.0000000000003875. PMID 27336874
- [Background] Kumagai Y, Ishiguro T, Haga N, Kuwabara K, Kawano T, Ishida H. Hemodynamics of the reconstructed gastric tube during esophagectomy: assessment of outcomes with indocyanine green fluorescence. World J Surg. 2014 Jan;38(1):138-43. doi: 10.1007/s00268-013-2237-9. PMID 24196170
- [Background] Yamaguchi K, Kumagai Y, Saito K, Hoshino A, Tokairin Y, Kawada K, Nakajima Y, Yamazaki S, Ishida H, Kinugasa Y. The evaluation of the gastric tube blood flow by indocyanine green fluorescence angiography during esophagectomy: a multicenter prospective study. Gen Thorac Cardiovasc Surg. 2021 Jul;69(7):1118-1124. doi: 10.1007/s11748-021-01640-2. Epub 2021 Apr 30. PMID 33929678